CLINICAL TRIAL: NCT01096030
Title: Uncontrolled, Open-label, Non-randomized, Phase 1 Study to Investigate the Pharmacokinetics, Safety, Tolerability, and Efficacy of BAY73-4506 in Chinese Patients With Advanced, Refractory Solid Tumors
Brief Title: Phase I Study of BAY73-4506 in Chinese Patients With Advanced, Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14996
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Neoplasms
Keywords: Regorafenib; Advanced; Refractory solid tumors
MeSH Terms: conditions — Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Experimental)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — 160 mg oral once daily BAY 73-4506 for 3 weeks of every 4 week cycle (i.e. 3 weeks on, 1 week off)

SUMMARY:
This will be an uncontrolled, open-label, non-randomized, phase I study. The primary objectives of this study are to define the pharmacokinetics (PK) and to evaluate the safety and tolerability of Regorafenib administered orally as a single agent in Chinese patients with advanced solid tumors. The secondary objectives are to evaluate tumor response of patients treated with Regorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese subjects >/- 18 years
* Advanced, histologically or cytologically confirmed solid tumors
* Subjects malignancies must be refractory to standard treatment or have no standard therapy available, or the subject actively refused any treatment that would be regarded standard, and/or if, in the judgment of the investigator or his/her designated associate(s), experimental treatment is clinically and ethically acceptable.
* Eastern Cooperative Oncology Group performance status (ECOG-PS) 0-1;
* Adequate bone marrow, liver and renal function
* Life expectancy of at least 3 months

Exclusion Criteria:

* Unstable/uncontrolled cardiac disease
* History of arterial or venous thrombotic or embolic events
* Malabsorption condition
* Severe renal impairment; persistent proteinuria >/= Grade 3
* Symptomatic metastatic brain or meningeal tumors
* Clinically significant bleeding >/=Grade 3 within 30 days before start of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics as measured by cmax and AUC | Cycle 0, Day 1-5,Cycle 1 Day 1,8,15,21,Cycle 2 Day 1,Modified Dosing Cycle Day 21
Adverse Event collection | every 1-2 weeks

SECONDARY OUTCOMES:
Objective tumor response rate | Every 8 weeks for the first 6 cycles, afterwards every 12 weeks

OTHER OUTCOMES:
Exploratory biomarker analysis | Screening, Cycle 0 or 1

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Hong Kong (2):
  - Shatin, N.T
  - Hong Kong
- Singapore, Singapore